CLINICAL TRIAL: NCT05896644
Title: An Evaluation of Eat Well, a Produce Benefit, for Patients With Diabetes and At-risk for Food Insecurity
Brief Title: Eat Well Produce Benefit for Diabetes and Food Insecurity
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00112649
Record Dates: First submitted 2023-05-26; First posted 2023-06-09 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Diabetes Mellitus; Food Insecurity
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eat Well (Experimental): The experimental group will participate in the Eat Well Produce Prescription program, receiving an $80 monthly benefit for eligible produce for 12 months and diabetes education materials through email, including curated nutrition and diet information from the Diabetes Resource Page, consistent with standard of care at Duke University Health System.
  Interventions: Other: Eat Well
- Control (No Intervention): The control group will receive usual care (including diabetes educational materials) without the prescription benefit.

INTERVENTIONS:
Other: Eat Well — A program offered by Reinvestment Partners giving clients gift/debit cards that allow the purchase of WIC approved fruits and vegetables.
  Arms: Eat Well

SUMMARY:
The goal of this clinical trial is to assess the impact of participation in Eat Well for diabetes patients who are at risk of food insecurity. The main questions it aims to answer are:

* whether there is a difference in Haemoglobin (Hb) A1c measurements and emergency department (ED) utilization between the Eat Well and control groups up to 18 months post-program completion.
* whether there are differences in cardiometabolic health-related outcomes for Eat Well participants.

Participants in the program will receive gift/debit cards for fruits and vegetables and educational nutrition materials. Researchers will compare Eat Well participants with those only receiving educational materials to see if there are differences in cardiometabolic health outcomes.

DETAILED DESCRIPTION:
This pragmatic trial aims to assess the impact of Eat Well participation for diabetes patients at risk of food insecurity. Eligible patients will receive gift/debit cards for the Special Supplemental Nutrition Program for Women, Infants, and Children (WIC)-approved fruits and vegetables and be assigned to either receive the card for up to 12 months or not. Random assignment will occur using a 2 to 1 treatment to control allocation ratio. Both treatment and control groups will receive curated diabetes educational materials. The study will assess the impact of the intervention on clinical factors such as glycemic control, weight, BMI, lipids, medication adherence, medication number, blood pressure, and utilization up to 18 months pre, during, and post program enrollment using data from clinical visits. The primary analysis of interest will be differences in HbA1c measurements and ED visits between the Eat Well and control groups at 12 months of program participation, with further evaluation of differences at 12 months post-program completion.

ELIGIBILITY:
Inclusion Criteria:

* Be active in the Duke Diabetes Registry in the past 12 months AND
* have had at least one outpatient A1c measurement AND
* are at risk for food insecurity as defined by one of the following:

  1. answered often true or sometimes true on one or both of the food insecurity questions as part of the electronic health record social history section (Maestro Care/ Epic of Verona WI) OR
  2. answered hard or very hard to the financial stress question as part of the electronic health record social history section (Maestro Care/ Epic of Verona WI) OR
  3. has Medicaid as insurance payer OR
  4. lives in Area Deprivation Index (ADI) zip code of 7th decile or harder

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2177 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2024-07-16 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1C | 18 months pre program, during program enrollment, up to 12 months
  A measure of average blood sugar levels over the past 3 months.
Change in number of ED Visits | up to 18 months pre program, during program enrollment, up to 12 months
  Number of ED visits throughout the study period

SECONDARY OUTCOMES:
Outpatient visits | up to 18 months pre program, during program, and up to 18 months post program
  Number of outpatient visits during the study period
Hospitalizations | up to 18 months pre program, during program, and up to 18 months post program
  Number of patient hospitalizations during the study period
Change in weight | up to 18 months pre program, during program, and up to 18 months post program enrollment
Change in body mass index (BMI) | up to 18 months pre program, during program, and up to 18 months post program
  A measure of body fat based on height and weight.
Change in cholesterol | up to 18 months pre program, during program, and up to 18 months post program
  Measure of lipids
Medication adherence (proportion of days covered) | up to 18 months pre program, during program, and up to 18 months post program
  Medication adherence will be measured by linking EHR data with Surescripts e-prescription network data. Surescripts facilitates medication refill information exchange between healthcare organizations and pharmacies. Adherence will be calculated using the proportion of days covered (PDC) approach
Change in number of diabetes and hypertension medications | up to 18 months pre program, during program, and up to 18 months post program
  Change in diabetes and hypertension medication numbers
Change in blood pressure | up to 18 months pre program, during program, and up to 18 months post program
  Systolic and Diastolic blood pressure
Change in HbA1C | 18 months post program
  A measure of average blood sugar levels over the past 3 months.
Change in number of ED Visits | 18 months post program
  Number of ED visits throughout the study period

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Access to all participant data and information will be restricted to authorized personnel. Internal monitoring of data may occur as required by Duke for investigator-initiated clinical research.

REFERENCES:
- [Derived] Drake C, Granados I, Rader A, Brucker A, Hoeffler S, Goldstein BA, Chamorro C, Johnson F, Hinz EM, Bedoya AD, German JC, Hauser J, Thacker C, Spratt SE. Addressing cost barriers to healthy eating with Eat Well, a prescription produce subsidy, for patients with diabetes and at risk for food insecurity: Study protocol for a type 1 hybrid effectiveness-implementation pragmatic randomized controlled trial. Contemp Clin Trials. 2024 Oct;145:107655. doi: 10.1016/j.cct.2024.107655. Epub 2024 Aug 5. PMID 39111387
- See also: Resource guide to be provided to all patients, regardless of selection in intervention or control group — http://diabetes.my.dukehealth.org
- See also: Link provided to all patients to find diabetes self management education and support in their area — https://nf01.diabeteseducator.org/eweb/DynamicPage.aspx?Site=aade&WebCode=DEAPFindApprovedProgram